CLINICAL TRIAL: NCT01331005
Title: A Phase II Evaluation of Topical Non-steroidal Anti-inflammatories in Eyes With Non Central Involved Diabetic Macular Edema
Brief Title: NSAID Phase II for Non-central Involved Diabetic Macular Edema (DME)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRCR.net Protocol R; U10EY018817-03 (NIH); U10EY014231-09 (NIH)
Record Dates: First submitted 2011-04-06; First posted 2011-04-07 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Macular Edema
Keywords: Macular Edema; Non steroidal anti-inflammatories
MeSH Terms: conditions — Macular Edema | interventions — nepafenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be given three times per day for one year
  Interventions: Other: Nepafenac Vehicle
- nepafenac 0.1% drops (Active Comparator): Nepafenac drops will be given three times per day for one year
  Interventions: Drug: nepafenac 0.1% drops

INTERVENTIONS:
Drug: nepafenac 0.1% drops — One drop three times per day for one year
  Arms: nepafenac 0.1% drops
Other: Nepafenac Vehicle — Placebo
  Arms: Placebo

SUMMARY:
This study is being conducted to assess the effects of topical nonsteroidal anti-inflammatories (NSAIDs) on macular retinal volume compared with placebo in eyes with non-central diabetic macular edema (DME). A secondary objective of this study is to assess the effects of topical NSAIDs on central subfield thickness and to compare the progression of non-central DME to central DME as determined by optical coherence tomography (OCT) and stereoscopic fundus photographs. Furthermore, this phase II study is being conducted (1) to determine whether the conduct of a phase III trial has merit based on an anatomic outcome, (2) to estimate recruitment potential of a phase III investigation, and (3) to provide information on outcome measures needed to design a phase III trial. The study is not designed to establish the efficacy of NSAIDs in the treatment of non- central DME.

DETAILED DESCRIPTION:
There is strong evidence to indicate that prevention of non-central involved DME from progression into the central subfield of the macula is a good anatomic surrogate for preventing visual acuity loss. Furthermore, the prevalence of macular edema is estimated to be high among patients with diabetes, and it is likely that approximately 25% of non-central involved cases of DME extend into the central subfield of the macula within one year. Thus, if a relatively safe and economical treatment could be identified that reduced the progression of non-central involved edema to central-involved edema by at least 50%, this treatment could have a major public health impact.

There is also evidence that inflammation has a role in DME, and that a topical NSAID might have an effect on retinal edema. Topical NSAIDs are in current widespread clinical use and appear to be well tolerated and safe when administered chronically, making them a potentially attractive alternative treatment for DME in patients who would like to delay or avoid laser photocoagulation or intravitreal injections (for example, patients who are willing to use daily eye drops to avoid ocular procedures or patients for whom access to experienced retinal specialists to apply laser photocoagulation or other treatments is limited).

This phase II trial may provide proof of concept evidence that topical NSAID treatment can have a beneficial effect on DME and possibly prevent increases in retinal volume or progression of non central-involved DME into the central subfield of the macula. Furthermore, it could determine the correlation between OCT and fundus photographic documentation of progression of DME into the central subfield in this clinical trial setting. Since effective treatments, including laser photocoagulation and intravitreal injections, already exist for DME treatment, topical NSAIDs would have to demonstrate a substantial effect on DME progression in order to be of sufficient clinical interest for further investigation. If a beneficial effect is apparent in this trial, which utilizes a relatively small sample size and short follow-up period, results from this phase II study might be utilized in planning future phase III trials. These future phase III trials could definitively answer whether or not NSAIDs are an efficacious novel therapeutic approach to the treatment of DME or preventing the progression of DME from extending into the central subfield of the macula.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Type 1 or type 2 diabetes
* Only one study eye per subject may be enrolled. The study eye must meet the following:

  * Best corrected E-ETDRS visual acuity letter score ≥ 74 (i.e., 20/32 or better) within 8 days of enrollment.
  * On clinical exam, definite retinal thickening due to DME within 3000 μm of the center of the macula but not involving the central subfield.
  * Thickened non-central macular subfields on DRCR.net approved spectral domain OCT macular map.
  * Central subfield thickness within threshold definition for normal central subfield thickness on DRCR.net approved spectral domain OCT machine.
  * No focal/grid laser within the last 6 months or other treatment for DME within the last 4 months.
  * No anticipated need to treat DME during the course of the study, unless the eye meets the criteria for treatment (Central subfield retinal thickness increases to 310 μm or more in spectral domain OCT machine from baseline).
* Diagnosis of diabetes mellitus (type 1 or type 2). Any one of the following will be considered to be sufficient evidence that diabetes is present:

  * Current regular use of insulin for the treatment of diabetes.
  * Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes.
  * Documented diabetes by American Diabetes Association and/or the World Health Organization criteria.
* At least one eye meets the study eye criteria.
* Able and willing to provide informed consent.
* Successful completion of the run-in phase during which level of compliance is more than 80%

Study Eye Inclusion Criteria

* Best corrected E-ETDRS visual acuity letter score ≥74 (i.e.20/32 or better) within 8 days of randomization.
* On clinical exam, definite retinal thickening due to DME within 3000 μm of the center of the macula but not involving the central subfield.
* Thickened non-central macular subfields on spectral domain OCT macular map that meet either of the following criteria:

  * At least two non-central macular subfields with OCT thickness above threshold (average normal + 2 SD) from DRCR.net approved spectral domain OCT machines- see below.
  * At least one non-central macular subfield with OCT thickness at least 15 μm above threshold (average normal + 2 SD) from DRCR.net approved spectral domain OCT machines-see DRCR.net procedures manual for threshold details.
* Central subfield thickness <250 microns obtained by one of the following DRCR.net approved spectral domain OCT machines:

  * Zeiss Cirrus
  * Heidelberg Spectralis
  * Optovue RTVue
* Media clarity, pupillary dilation, and study participant cooperation sufficient for adequate OCT and fundus photographs.
* If the study participant is on multiple ocular drops, investigator believes that study participant can be compliant with a multi-drop regimen.

Exclusion Criteria:

A study participant is not eligible for the run-in phase or the randomized trial if any of the following exclusion criteria are present:

* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Subjects in poor glycemic control who, within the last 4 months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 4 months should not be enrolled.
* Use of systemic corticosteroids or anti-VEGF therapy.
* Current use of prescription systemic NSAIDs.
* History of auto-immune diseases such as rheumatoid arthritis.
* Participation in an investigational trial that involved treatment with any drug within 30 days of randomization that has not received regulatory approval at the time of study entry.
* Note: study participants cannot receive another investigational drug while participating in the study.
* Known allergy to any component of the study drug.
* Blood pressure > 180/110 mmHg (systolic above 180 or diastolic above 110 mmHg)
* If blood pressure is brought below 180/110 by anti-hypertensive treatment, study participant can become eligible.
* Participant is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the 12 months of the study.
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 12 months.
* Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgment is used to determine when a pregnancy test is needed.

Study Eye Exclusion Criteria

* History of focal/grid laser within the last 6 months or other treatment for DME within the last 4 months

  -Note: Throughout the study, the distribution of subjects with prior treatment for DME will be evaluated, and eligibility criteria may be tailored to add balance between subjects with prior treatment and subjects without prior treatment for DME.
* Anticipated need to treat DME during the course of the study (Any DME treatment during the study should follow criteria in section 4.3).
* History of use of NSAID eye drops within the last 30 days or anticipated need for such drops during the study due to other ocular condition
* History of panretinal (scatter) photocoagulation (PRP) within 4 months prior to randomization
* Anticipated need for PRP in the 6 months following randomization
* Anticipated need for cataract extraction surgery in the study eye during the study period
* Lipid in the fovea (center of the macula)
* History of major ocular surgery (including scleral buckle, any intraocular surgery, etc.) within prior 4 months or major ocular surgery anticipated within the next 6 months following randomization
* An ocular condition, other than diabetic macular edema, is present such that, in the opinion of the investigator, visual acuity might be affected now (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, non-retinal condition, epiretinal membrane or vitreo-macular traction) or during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.)
* History of YAG capsulotomy performed within 2 months prior to randomization
* Exam evidence of severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis
* Aphakia
* History of vitrectomy for any reason
* History of cataract surgery within the prior 1 year
* Uncontrolled glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Friedman, MD, Principal Investigator — Florida Retina Consultants
Locations (32):
- United States (32):
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Southern California Desert Retina Consultants, MC, Palm Springs, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retinal Consultants of Southern California Medical Group, Inc., Westlake Village, California
  - Retina Consultants of Southwest Florida, Fort Myers, Florida
  - Central Florida Retina Institute, Lakeland, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Retina Associates of Hawaii, Inc., Honolulu, Hawaii
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - American Eye Institute, New Albany, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina and Vitreous Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Henry Ford Health System, Dept of Ophthalmology and Eye Care Services, Detroit, Michigan
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Eyesight Ophthalmic Services, PA, Portsmouth, New Hampshire
  - Eye Care for the Adirondacks, Plattsburgh, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - Charlotte Eye Ear Nose and Throat Assoc, PA, Charlotte, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Retina Northwest, PC, Portland, Oregon
  - Family Eye Group, Lancaster, Pennsylvania
  - Southeastern Retina Associates, PC, Kingsport, Tennessee
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Texas Retina Associates, Lubbock, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Friedman SM, Almukhtar TH, Baker CW, Glassman AR, Elman MJ, Bressler NM, Maker MP, Jampol LM, Melia M; Diabetic Retinopathy Clinical Research Network. Topical nepafenec in eyes with noncentral diabetic macular edema. Retina. 2015 May;35(5):944-56. doi: 10.1097/IAE.0000000000000403. PMID 25602634

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Nepafenac 0.1% Drops
Started | 64 | 61
Completed | 60 | 57
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nepafenac 0.1% Drops | Total
Number analyzed (Participants) | 64 | 61 | 125
Age, Customized [Median (Inter-Quartile Range); unit: years] | 59 [51 to 66] | 60 [52 to 68] | 60 [51 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 36 | 38 | 74
Race/Ethnicity, Customized [Number; unit: participants]
  White | 38 | 44 | 82
  African American | 13 | 7 | 20
  Hispanic or Latino | 12 | 5 | 17
  American Indian/Alaskan Native | 1 | 0 | 1
  Native Hawaiian/Other Pacific Islander | 0 | 2 | 2
  Asian | 0 | 2 | 2
  More than one race | 0 | 1 | 1
Type of Diabetes [Number; unit: participants]
  Type 1 | 5 | 5 | 10
  Type 2 | 56 | 53 | 109
  Uncertain | 3 | 3 | 6
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 17 (11) | 19 (11) | 18 (11)
Hemoglobin A1c [Median (Inter-Quartile Range); unit: Percent HbA1c] | 7.9 [7.2 to 10] | 8.1 [7.1 to 8.7] | 7.9 [7.1 to 9.0]
Electronic-Early Treatment Diabetic Retinopathy Study Visual Acuity Letter Score [Mean (Standard Deviation); unit: units on a scale] — Visual acuity was measured with the E-ETDRS method and resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
  units on a scale | 83 (7) | 82 (6) | 83 (7)
History of Diabetic Macular Edema Treatment [Number; unit: participants]
  yes | 28 | 30 | 58
  no | 36 | 31 | 67
History of Panretinal Photocoagulation [Number; unit: participants]
  yes | 11 | 13 | 24
  no | 53 | 48 | 101
Optical Coherence Tomography Machine [Number; unit: participants]
  Zeiss Cirrus | 41 | 37 | 78
  Heidelberg Spectralis | 23 | 24 | 47
Optical Coherence Tomography Central Subfield Thickness [Mean (Standard Deviation); unit: Microns] | 218 (25) | 227 (29) | 223 (27)
Optical Coherence Tomography Retinal Volume [Mean (Standard Deviation); unit: mm^3] | 7.7 (0.4) | 7.9 (0.6) | 7.8 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Optical Coherence Tomography Measure Retinal Volume, mm3
Time Frame: From Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: mm3
Arm/Group | Placebo | Nepafenac 0.1% Drops
Number analyzed (Participants) | 64 | 61
mm3 | 0.02 [-0.19 to 0.16] | -0.03 [-0.21 to 0.14]

2. Secondary Outcome: Mean Change in Visual Acuity
Description: Visual Acuity was measured with the Electronic Early Treatment Study (E-ETDRS) visual acuity test. Unit of measure is based on the E-ETDRS letter score scale, 0-97, where 0 = worst and 97 = best.
Time Frame: baseline to 12 months
Population: Original 12-month values are not available in 4 eyes of each of nepafenac and placebo groups because 12-month visit was not completed and were imputed from the last available measurement; values at or before first diabetic macular edema treatment were carried forward in 5 and 3 eyes of nepafenac and placebo groups respectively.
Measure: Mean (Standard Deviation); unit: Letter Score
Arm/Group | Placebo | Nepafenac 0.1% Drops
Number analyzed (Participants) | 64 | 61
Letter Score | -0.3 (6.2) | 0.2 (5.7)

3. Secondary Outcome: Change in OCT Central Subfield Thickness
Description: 95% CI will be obtained in each treatment group and compared between treatment groups at 1 year. For eyes that have received treatment for DME before 1 year, visual acuity and OCT measurements obtained at time of failure will be used instead of measurements at 1 year.
Time Frame: baseline to 12 months
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Placebo | Nepafenac 0.1% Drops
Number analyzed (Participants) | 64 | 61
microns | 7 (35) | 9 (45)

ADVERSE EVENTS:
Arm/Group | Placebo | Nepafenac 0.1% Drops
Serious Adverse Events (participants affected / at risk) | 12/64 | 16/61
Other Adverse Events (participants affected / at risk) | 37/64 | 30/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | Nepafenac 0.1% Drops (N=61)
Burning Eyes (Eye disorders) | 0 (0) | 1 (1)
Chemical Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Corneal Melt (Eye disorders) | 0 (0) | 1 (1)
Vision Decreased (Eye disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Bowl Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 2 (2) | 1 (1)
Gallbladder Stones (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shoulder Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Kidney Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Spinal stenosis of unspecified region (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (cerebrovascular accident) (Nervous system disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Gastric bypass surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Removal of foreign body from throat (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Caratoid artery disease (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | Nepafenac 0.1% Drops (N=61)
Eye Pain (Eye disorders) | 5 (5) | 1 (1)
Blurred Vision (Eye disorders) | 6 (6) | 6 (6)
Floaters (Eye disorders) | 4 (4) | 4 (4)
Vitreous Hemorrhage (Eye disorders) | 1 (1) | 4 (4)
Cataract (Eye disorders) | 3 (3) | 3 (3)
Chest Pain (Cardiac disorders) | 3 (3) | 2 (2)
Eye Itching (Eye disorders) | 3 (3) | 0 (0)
Fall (General disorders) | 3 (3) | 1 (1)
Proliferative Diabetic Retinopathy (Eye disorders) | 3 (3) | 0 (0)
Stomach Virus (Gastrointestinal disorders) | 2 (2) | 3 (3)
Vision Decreased (Eye disorders) | 3 (3) | 3 (3)
Visual Acuity Decreased (Eye disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Members of the Network can not discuss the trial results until the primary outcome has been made publicly available.